CLINICAL TRIAL: NCT06979271
Title: Clinical Efficacy and Safety of Real-world Patients With Refractory Rheumatoid Arthritis (D2TRA) Receiving Telitacicept in Combination With Tofacitinib
Brief Title: Efficacy and Safety of Telitacicept Combined With Tofacitinib for Refractory Rheumatoid Arthritis
Status: Recruiting | Type: Observational
Sponsor: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Zhenhua Ying, Director, Zhejiang Provincial People's Hospital
Other Study IDs: KT2025024
Record Dates: First submitted 2025-05-06; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Telitacicept; Treatment Compliance; Rheumatoid Arthritis
MeSH Terms: conditions — Patient Compliance; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Telitacicept Tofacitinib — One group of D2TRA subjects receive Telitacicept combine Tofacitinib treatment

SUMMARY:
The aim of this study is to observe the clinical efficacy and safety of telitacicept combined with tofacitinib in the treatment of D2TRA patients

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-85 years
2. Diagnosed with refractory rheumatoid arthritis according to the 2021 EULAR (European Alliance of Associations for Rheumatology) diagnostic criteria
3. The traditional disease-improving rheumatic drug treatment is ineffective, and the use of two or more biological/targeted disease-improving anti-rheumatic drugs is ineffective, and telitacicept combined with tofacitinib is required treated patients
4. Voluntarily provided written informed consent -

Exclusion Criteria:

1. Exclusion of patients with severe diseases of major organs (e.g., heart, liver, or lungs)
2. Patients with malignancies, hematological disorders, or other autoimmune diseases (excluding rheumatoid arthritis)
3. History of allergy/hypersensitivity to the study medications (Telitacicept or Tofacitinib)
4. Active tuberculosis or active infectious diseases requiring systemic treatment
5. Pregnancy, lactation, or refusal to use contraception during the study
6. Failure to complete the prescribed Telitacicept + Tofacitinib regimen due to: Non-adherence or Severe adverse reactions
7. Other conditions contraindicating participation per investigator judgment -

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with refractory rheumatoid arthritis
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Telitacicept Combined With Tofacitinib for Refractory Rheumatoid Arthritis | maximum 1 years
  The disease activity score of 28 joints with erythrocyte sedimentation rate (DAS28-ESR ≤ 2.6, remission; 2.6 < DAS28-ESR ≤ 3.2, mild activity; 3.2 < DAS28-ESR ≤ 5.1, moderate activity, and DAS28-ESR > 5.1, severe activity)

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse EventsArthritis | maximum 1 years
  Liver and kidney function

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
No plan to share data

REFERENCES:
- [Result] Zeng L, Yang K, Wu Y, Yu G, Yan Y, Hao M, Song T, Li Y, Chen J, Sun L. Telitacicept: A novel horizon in targeting autoimmunity and rheumatic diseases. J Autoimmun. 2024 Sep;148:103291. doi: 10.1016/j.jaut.2024.103291. Epub 2024 Aug 14. PMID 39146891

DOCUMENTS (2):
  • Study Protocol (2025-04-09): https://cdn.clinicaltrials.gov/large-docs/71/NCT06979271/Prot_000.pdf
  • Informed Consent Form (2025-04-09): https://cdn.clinicaltrials.gov/large-docs/71/NCT06979271/ICF_001.pdf